CLINICAL TRIAL: NCT04401267
Title: Hypertension Intervention to Reduce Osteonecrosis in Children With Acute Lymphoblastic Leukemia/Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HYPERION; 1K08CA250418 (NIH); NCI-2020-03603 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2020-05-13; First posted 2020-05-26 (Actual); Results first posted 2024-07-11 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Hypertension; Osteonecrosis; Osteonecrosis Due to Drug
Keywords: Acute Lymphoblastic Leukemia; Children; Hypertension; Osteonecrosis; Osteonecrosis Due to Drug
MeSH Terms: conditions — Hypertension; Osteonecrosis; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Evaluation of the MRIs defining the primary endpoint will be performed by a blinded radiologist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intensive Antihypertensive Therapy (Experimental): Patients will begin Intensive antihypertensive therapy to achieve the targeted blood pressure (targeted to the 50-75th percentile for age, sex, and height) on day 4 of Remission Induction on TOT17 and continue during steroid containing phases until the completion of reinduction II.
  Interventions: Drug: Intensive Antihypertensive Therapy; Other: Symptom Survey; Other: Semi-structured interview
- Conventional Antihypertensive Therapy (Active Comparator): Patients will begin Conventional antihypertensive therapy to achieve the targeted blood pressure (targeted to the 90-95th percentile for age, sex, and height) on day 4 of Remission Induction on TOT17 and continue during steroid containing phases until the completion of reinduction II.
  Interventions: Drug: Conventional Antihypertensive Therapy; Other: Symptom Survey; Other: Semi-structured interview

INTERVENTIONS:
Drug: Intensive Antihypertensive Therapy — Receives intensive antihypertensive therapy
  Other Names: Hypotensive Therapy
  Arms: Intensive Antihypertensive Therapy
Drug: Conventional Antihypertensive Therapy — Receives conventional antihypertensive therapy
  Other Names: Hypotensive Therapy
  Arms: Conventional Antihypertensive Therapy
Other: Symptom Survey — The symptom survey is comprised of the PROMIS Ped 25 profile, PROMIS pain interference 8a, PROMIS physical activity 8a, and PROMIS mobility 8a during induction (day 23-28), during week 17 of continuation (+/- 2 weeks), and continuation week 49 (+/- 3 weeks).
  Other Names: Survey
Other: Semi-structured interview — Patients will be interviewed by a trained examiner about their treatment and symptom burden on Week 49 of TOT17 Continuation Therapy. The interview will be recorded and will take about 30-45 minutes.
  Other Names: Interview

SUMMARY:
This is a randomized unblinded Phase II clinical trial evaluating the impact of intensive antihypertensive control (targeted to the 50-75th percentile for age, sex, and height) compared to conventional antihypertensive control (targeted to the 90-95th percentile for age, sex, and height) on the incidence of radiographically extensive osteonecrosis in children and young adults receiving treatment for newly diagnosed acute lymphoblastic leukemia/lymphoma (ALL).

Primary Objective

* Compare the frequency of radiographically extensive osteonecrosis in patients receiving intensive compared to conventional antihypertensive therapy.

Secondary Objectives

* Evaluate the efficacy of intensive antihypertensive control compared to conventional antihypertensive control in the prevention of clinically significant (CTCAE Grade 2 or higher) and radiologically extensive osteonecrosis, overall and stratified by joints.
* Compare the frequency of clinically significant and radiographically extensive osteonecrosis in patients receiving antihypertensive therapy and historical controls.
* Compare blood pressures achieved in intensive and conventional arms using both pressures obtained as part of routine patient care and ambulatory blood pressure monitoring.
* Compare levels of vascular dysfunction as measured physiologically, radiographically, and in blood samples in patients receiving intensive compared to standard antihypertensive therapy.

Exploratory Objectives

* Identify predictive patterns of blood biomarkers which identify patients at high- risk of developing clinically significant osteonecrosis.
* Identify MRI findings during late induction which correlate with osteonecrosis lesions seen during reinduction.
* Identify patterns of diurnal blood pressure variation as measured by ambulatory blood pressure monitoring associated with the later development of osteonecrosis.
* Compare induction blood pressure control and intervention arm to echocardiographic changes at reinduction II.
* Evaluate patient-reported, health-related quality of life in patients during induction and after 1.5 years of therapy when many experience the symptoms of osteonecrosis.

DETAILED DESCRIPTION:
Patient randomization will be stratified based on patient's location (Memphis vs. other), use of antihypertensives prior to randomization, and factors known to influence osteonecrosis risk, specifically sex and self-declared race (non-Hispanic white vs. other). A target systolic blood pressure range will be chosen for each participant based on their randomization arm, age, sex, and height.

Patients will be randomized on day 4 of induction therapy to either conventional or intensive blood pressure goals. Patients will be treated with antihypertensive therapy to achieve blood pressure control as indicated by their randomized arm. Therapy will be adjusted every 3-4 days as needed to achieve targeted control based on the mean of blood pressures obtained in that period. Treatment of hypertension to the target will continue until the completion of reinduction II therapy. Patients will be evaluated for osteonecrosis as indicated in their primary therapeutic protocol using MRI during reinduction II.

Patients will be asked to complete a symptom survey and a semi-structured interview.

ELIGIBILITY:
Inclusion Criteria:

* Patient is being treated for newly diagnosed acute lymphoblastic leukemia or lymphoma (ALL) on the TOT17 protocol. Patients do not need to be hypertensive to enroll.
* Patient is 10 years of age or older at the time of enrollment on TOT17.
* Patient has completed ≤ 4 days of protocol therapy (patients are eligible on Day 4 of TOT17 therapy).

Exclusion Criteria:

* Moderate-severe renal dysfunction (glomerular filtration rate <45 ml/min/1.73m2).
* Down's syndrome (germline Trisomy 21) or other syndrome resulting in growth delay or alterations in stature.
* Chronic inability to ambulate. Patients with limitations in movement due to acute complications of leukemia/lymphoma are not excluded.
* Permanent contraindication to MRI evaluation.
* Participants who are pregnant or lactating. Males or females of reproductive potential must agree to use effective contraception for the duration of study participation.
* Inability or unwillingness of research participant or legal guardian/representative to give written informed consent.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2023-09-25 (Actual); Study Completion 2025-10-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Seth E. Karol, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (2):
- United States (2):
  - St. Jude Affiliate Clinic - Novant Health Hemby Children's Hospital, Charlotte, North Carolina
  - St. Jude Children's Research Hospital, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Individual participant de-identified datasets containing the variables analyzed in the published article will be made available (related to the study primary or secondary objectives contained in the publication). Supporting documents such as the protocol, statistical analyses plan, and informed consent are available through the CTG website for the specific study. Data used to generate the published article will be made available at the time of article publication. Investigators who seek access to individual level de-identified data will contact the computing team in the Department of Biostatistics (ClinTrialDataRequest@stjude.org) who will respond to the data request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available at the time of article publication.
Access Criteria: Data will be provided to researchers following a formal request with the following information: full name of requestor, affiliation, data set requested, and timing of when data is needed. As an informational point, the lead statistician and study principal investigator will be informed that primary results datasets have been requested.

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: ClinicalTrials Open at St. Jude — http://www.stjude.org/protocols

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 51 patients were enrolled into the study from 15OCT2020 to 28DEC2022. Of those, one patient was found to be ineligible to the study. Therefore, only 50 eligible patients will be included in the analyses of the study.
Groups:
- Conventional (Standard) Antihypertensive Therapy: Patients will begin Conventional antihypertensive therapy to achieve the targeted blood pressure (targeted to the 90-95th percentile for age, sex, and height) on day 4 of Remission Induction on TOT17 and continue during steroid containing phases until the completion of reinduction II.
Period: Overall Study
Arm/Group | Intensive Antihypertensive Therapy | Conventional (Standard) Antihypertensive Therapy
Started | 26 | 25
Completed | 21 | 22
Not Completed | 5 | 3
Not completed — Death | 0 | 1
Not completed — Discontinuation of TOT17 therapy | 4 | 2
Not completed — Found to be Ineligible | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Conventional (Standard) Antihypertensive Therapy | Intensive Antihypertensive Therapy | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.96 (1.86) | 14.27 (2.42) | 14.11 (2.14)
Age, Continuous [Median (Full Range); unit: years] | 13.93 [10.58 to 18.54] | 14.01 [10.07 to 18.43] | 13.98 [10.07 to 18.54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 16 | 15 | 31
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 13 | 16 | 29
  Black | 7 | 6 | 13
  Other | 4 | 1 | 5
  Missing | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Extensive Radiographic Osteonecrosis
Description: Involvement of >=30% of the epiphyseal surface of either the hip or knee by prospective MRI during reinduction II
Time Frame: during reinduction II therapy, approximately 9 months into therapy.
Population: There were 21 of the 25 patients in conventional group, and 23 of the 25 patients in Intensive group reached reinduction II and had the MRI measurement during reinduction II.
Measure: Count of Participants; unit: Participants
Arm/Group | Conventional (Standard) Antihypertensive Therapy | Intensive Antihypertensive Therapy
Number analyzed (Participants) | 21 | 23
Participants
  <30% | 20 | 21
  >=30% | 1 | 2
Statistical Analysis 1: Comparison: Conventional (Standard) Antihypertensive Therapy vs Intensive Antihypertensive Therapy; Test type: Superiority; p = 0.7139, Fisher Exact

2. Secondary Outcome: Rate of Clinically Significant Osteonecrosis
Description: CTCAE grade 2 or high osteonecrosis
Time Frame: any time during leukemia therapy, approximately 2.5 years
Reporting Status: Not Posted

3. Secondary Outcome: Rate of Clinically Significant Osteonecrosis vs. Historical Control
Description: CTCAE grade 2 or high osteonecrosis vs. Total 16 matched controls
Time Frame: any time during leukemia therapy, approximately 2.5 years
Reporting Status: Not Posted

4. Secondary Outcome: Blood Pressure Control on Trial
Description: Comparison of repeated systolic and diastolic blood pressure measures between randomized treatment arms
Time Frame: first 9 months of therapy
Population: Three patients on the Conventional Arm did not have the required measurement. Four patients on the Intensive Arm did not have the required measurement.
Measure: Median (Full Range); unit: mmHg
Arm/Group | Conventional (Standard) Antihypertensive Therapy | Intensive Antihypertensive Therapy
Number analyzed (Participants) | 22 | 21
mmHg
  Systolic Blood at Pressure at Month9 | 114.00 [103.00 to 127.00] | 117.00 [91.00 to 139.00]
  Diastolic Blood Pressure at Month9 | 70.00 [60.00 to 82.00] | 74.00 [54.00 to 87.00]

5. Secondary Outcome: Biomarkers of Vascular Dysfunction - eNO Synthetase (pg/mL)
Description: Comparison between randomized treatment arms
Time Frame: 3 weeks and 9 months into therapy
Population: Seven patients on the Conventional Arm and Intensive Arm, Week3, did not have the required measurement. Fourteen patients on the Conventional Arm and Intensive Arm, Month9, did not have the required measurement.
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Conventional (Standard) Antihypertensive Therapy | Intensive Antihypertensive Therapy
Number analyzed (Participants) | 18 | 18
pg/mL
  Week3 | 187.78 [12.68 to 2030.13] | 267.03 [11.87 to 226392.20]
  Month9: number analyzed (Participants) | 11 | 11
  Month9 | 193.28 [87.49 to 1096.74] | 266.53 [32.89 to 435387.25]

6. Secondary Outcome: Biomarker of Vascular Dysfunction - Von Willebrand Factor (%)
Description: Comparison between randomized treatment arms
Time Frame: 3 weeks and 9 months into therapy
Population: Nine patients on the Conventional Arm and 10 on the Intensive Arm, Week3, did not have the required measurement. Four patients on the Conventional Arm and Intensive Arm, Month9, did not have the required measurement.
Measure: Median (Full Range); unit: percentage (%)
Arm/Group | Conventional (Standard) Antihypertensive Therapy | Intensive Antihypertensive Therapy
Number analyzed (Participants) | 21 | 21
percentage (%)
  Week3: number analyzed (Participants) | 16 | 15
  Week3 | 195.00 [143.00 to 420.00] | 191.00 [118.00 to 420.00]
  Month9 | 211.00 [59.00 to 420.00] | 164.00 [82.00 to 352.00]

7. Secondary Outcome: Biomarker of Vascular Dysfunction - TNF-alpha (pg/mL)
Description: Comparison between randomized treatment arms
Time Frame: 3 weeks and 9 months into therapy
Population: One patient on the Conventional Arm and 2 patients on the Intensive Arm, Week3, did not have the required measurement. Five patients on the Conventional Arm and Intensive Arm, Month9, did not have the required measurement.
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Conventional (Standard) Antihypertensive Therapy | Intensive Antihypertensive Therapy
Number analyzed (Participants) | 24 | 23
pg/mL
  Week3 | 0.87 [0.25 to 1.73] | 0.79 [0.36 to 1.86]
  Month9: number analyzed (Participants) | 20 | 20
  Month9 | 1.56 [0.51 to 3.45] | 1.44 [0.41 to 26.32]

8. Secondary Outcome: Biomarker of Vascular Dysfunction - D-dimer (µg/mL)
Description: Comparison between randomized treatment arms
Time Frame: 3 weeks and 9 months into therapy
Population: Nine patients on the Conventional Arm and 8 patients on the Intensive Arm, Week3, did not have the required measurement. Four patients on the Conventional Arm and 5 patients on the Intensive Arm, Month9, did not have the required measurement.
Measure: Median (Full Range); unit: µg/mL
Arm/Group | Conventional (Standard) Antihypertensive Therapy | Intensive Antihypertensive Therapy
Number analyzed (Participants) | 21 | 20
µg/mL
  Week3: number analyzed (Participants) | 16 | 17
  Week3 | 0.85 [0.30 to 2.00] | 0.60 [0.27 to 2.77]
  Month9 | 0.44 [0.27 to 4.28] | 0.29 [0.27 to 1.10]

9. Secondary Outcome: Biomarker of Vascular Dysfunction - PAI-1 (AU/mL)
Description: Comparison between randomized treatment arms
Time Frame: 3 weeks and 9 months into therapy
Population: Nine patients on the Conventional Arm and the Intensive Arm, Week3, did not have the required measurement. Four patients on the Conventional Arm and 7 patients on the Intensive Arm, Month9, did not have the required measurement.
Measure: Median (Full Range); unit: AU/mL
Arm/Group | Conventional (Standard) Antihypertensive Therapy | Intensive Antihypertensive Therapy
Number analyzed (Participants) | 21 | 18
AU/mL
  Week3: number analyzed (Participants) | 16 | 16
  Week3 | 17.85 [2.00 to 293.00] | 15.80 [3.10 to 71.90]
  Month9 | 38.00 [2.00 to 100.00] | 41.10 [2.00 to 138.50]

10. Secondary Outcome: Biomarker of Vascular Dysfunction - E-selectin (ng/mL)
Description: Comparison between randomized treatment arms
Time Frame: 3 weeks and 9 months into therapy
Population: One patient on the Conventional Arm and 2 patients on the Intensive Arm, Week3, did not have the required measurement. Five patients on the Conventional Arm and the Intensive Arm, Month9, did not have the required measurement.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Conventional (Standard) Antihypertensive Therapy | Intensive Antihypertensive Therapy
Number analyzed (Participants) | 24 | 23
ng/mL
  Week3 | 23.53 [6.36 to 56.64] | 23.24 [8.30 to 100.14]
  Month9: number analyzed (Participants) | 20 | 20
  Month9 | 65.16 [19.37 to 144.30] | 53.68 [28.86 to 163.90]

11. Secondary Outcome: Biomarker of Vascular Dysfunction - ICAM-1 (ng/mL)
Description: Comparison between randomized treatment arms
Time Frame: 3 weeks and 9 months into therapy
Population: as for outcome 10
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Conventional (Standard) Antihypertensive Therapy | Intensive Antihypertensive Therapy
Number analyzed (Participants) | 24 | 23
ng/mL
  Week3 | 328.79 [166.05 to 515.52] | 314.22 [207.09 to 632.73]
  Month9: number analyzed (Participants) | 20 | 20
  Month9 | 629.13 [344.67 to 1620.85] | 639.25 [244.27 to 1511.56]

12. Secondary Outcome: Biomarker of Vascular Dysfunction - Arterial Elasticity (ml/mmHg)
Description: Comparison between randomized treatment arms
Time Frame: 3 weeks and 3 months into therapy
Population: Two patients on the Conventional Arm and Intensive Arm, Week3, did not have the required measurement. Seven patients on the Conventional Arm and 8 patients on the Intensive Arm, Month3, did not have the required measurement.
Measure: Median (Full Range); unit: ml/mmHg
Arm/Group | Conventional (Standard) Antihypertensive Therapy | Intensive Antihypertensive Therapy
Number analyzed (Participants) | 23 | 23
ml/mmHg
  Week3 | 11.60 [3.30 to 24.30] | 10.70 [3.00 to 21.00]
  Month3: number analyzed (Participants) | 18 | 17
  Month3 | 12.30 [6.80 to 18.80] | 10.40 [3.40 to 25.40]

13. Secondary Outcome: Biomarker of Vascular Dysfunction - Pulse Wave Velocity (m/Sec)
Description: Comparison between randomized treatment arms
Time Frame: 3 weeks and 3 months into therapy
Population: Two patients on the Conventional Arm and 3 patients on the Intensive Arm, Week3, did not have the required measurement. Eight patients on the Conventional Arm and on the Intensive Arm, Month3, did not have the required measurement.
Measure: Median (Full Range); unit: m/sec
Arm/Group | Conventional (Standard) Antihypertensive Therapy | Intensive Antihypertensive Therapy
Number analyzed (Participants) | 23 | 22
m/sec
  Week3 | 5.00 [0.50 to 8.30] | 5.35 [3.80 to 8.40]
  Month3: number analyzed (Participants) | 17 | 17
  Month3 | 5.00 [3.00 to 6.10] | 5.30 [3.10 to 6.10]

14. Secondary Outcome: Magnetic Resonance Imaging (MRI) of Right and Left Hip and Knee
Description: Comparison between randomized treatment arms on proportions of MRI identified lesions >= 30%.
Time Frame: 3 weeks and 9 months into therapy
Population: Four Conventional Arm patients and 2 Intensive Arm patients did not have Week3 right hip (R hip), left hip (L hip), right knee (R knee) and left knee (L knee) MRI.
  Five Conventional and Intensive Arm patients did not have Month9 R hip MRI. Four Conventional Arm patients and 5 Intensive Arm patients did not have a Month9 L hip and R knee MRI.
  Three Conventional Arm patients and 5 Intensive Arm patients did not have a Month9 L knee MRI.
Measure: Count of Participants; unit: Participants
Groups:
- Conventional (Standard) Antihypertensive Therapy-Magnetic Resonance Imaging (MRI)-Right Hip: Conventional (Standard) Antihypertensive Therapy-Magnetic resonance imaging (MRI) of Right Hip
- Intensive Antihypertensive Therapy-MRI-Right Hip: Intensive Antihypertensive Therapy-MRI of Right Hip
- Conventional (Standard) Antihypertensive Therapy-MRI-Left Hip: Conventional (Standard) Antihypertensive Therapy-MRI of Left Hip
- Intensive Antihypertensive Therapy-MRI-Left Hip: Intensive Antihypertensive Therapy-MRI of Left Hip
- Conventional (Standard) Antihypertensive Therapy-MRI-Right Knee: Conventional (Standard) Antihypertensive Therapy-MRI of Right Knee
- Intensive Antihypertensive Therapy-MRI-Right Knee: Intensive Antihypertensive Therapy-MRI of Right Knee
- Conventional (Standard) Antihypertensive Therapy-MRI-Left Knee: Conventional (Standard) Antihypertensive Therapy-MRI of Left Knee
- Intensive Antihypertensive Therapy-MRI-Left Knee: Intensive Antihypertensive Therapy-MRI of Left Knee
Arm/Group | Conventional (Standard) Antihypertensive Therapy-Magnetic Resonance Imaging (MRI)-Right Hip | Intensive Antihypertensive Therapy-MRI-Right Hip | Conventional (Standard) Antihypertensive Therapy-MRI-Left Hip | Intensive Antihypertensive Therapy-MRI-Left Hip | Conventional (Standard) Antihypertensive Therapy-MRI-Right Knee | Intensive Antihypertensive Therapy-MRI-Right Knee | Conventional (Standard) Antihypertensive Therapy-MRI-Left Knee | Intensive Antihypertensive Therapy-MRI-Left Knee
Number analyzed (Participants) | 21 | 23 | 21 | 23 | 21 | 23 | 22 | 23
Participants
  >=30% at Week3: number analyzed (Participants) | 21 | 23 | 21 | 23 | 21 | 23 | 21 | 23
  >=30% at Week3 | 1 | 2 | 1 | 2 | 1 | 1 | 1 | 1
  <30% at Week3: number analyzed (Participants) | 21 | 23 | 21 | 23 | 21 | 23 | 21 | 23
  <30% at Week3 | 20 | 21 | 20 | 21 | 20 | 22 | 20 | 22
  <30% at Month9: number analyzed (Participants) | 20 | 20 | 21 | 20 | 21 | 20 | 22 | 20
  <30% at Month9 | 17 | 16 | 18 | 16 | 18 | 16 | 19 | 16
  >=30% at Month9: number analyzed (Participants) | 20 | 20 | 21 | 20 | 21 | 20 | 22 | 20
  >=30% at Month9 | 3 | 4 | 3 | 4 | 3 | 4 | 3 | 4

ADVERSE EVENTS:
Time Frame: AEs will be collected approximately 9 months, until the end on reinduction.
Arm/Group | Intensive Antihypertensive Therapy | Conventional (Standard) Antihypertensive Therapy
All-Cause Mortality (participants affected / at risk) | 0/25 | 1/25
Serious Adverse Events (participants affected / at risk) | 22/25 | 22/25
Other Adverse Events (participants affected / at risk) | 24/25 | 24/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intensive Antihypertensive Therapy (N=25) | Conventional (Standard) Antihypertensive Therapy (N=25)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (6) | 9 (14)
Cardiac disorders - Other (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (2)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatic necrosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 4 (4) | 4 (4)
Vomiting (Gastrointestinal disorders) | 3 (3) | 2 (2)
Fever (General disorders) | 1 (1) | 1 (1)
Multi-organ failure (General disorders) | 0 (0) | 1 (1)
Allergic reaction (Immune system disorders) | 2 (2) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1) | 0 (0)
Eye infection (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Other (Infections and infestations) | 2 (2) | 3 (3)
Lung infection (Infections and infestations) | 2 (2) | 1 (1)
Mucosal infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 2 (4)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 2 (2) | 2 (3)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Blood antidiuretic hormone abnormal (Investigations) | 1 (1) | 2 (3)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 1 (1) | 1 (1)
Serum amylase increased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 4 (4)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 3 (3)
Syncope (Nervous system disorders) | 1 (1) | 1 (2)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
Mania (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 3 (3)
Renal calculi (Renal and urinary disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Hypotension (Vascular disorders) | 3 (4) | 4 (4)
Thromboembolic event (Vascular disorders) | 2 (2) | 2 (2)
Visceral arterial ischemia (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intensive Antihypertensive Therapy (N=25) | Conventional (Standard) Antihypertensive Therapy (N=25)
Alanine aminotransferase increased (Investigations) | 13 (33) | 13 (27)
Hyponatremia (Metabolism and nutrition disorders) | 10 (24) | 10 (20)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 13 (18) | 10 (17)
Hyperglycemia (Metabolism and nutrition disorders) | 6 (13) | 8 (12)
Mucositis oral (Gastrointestinal disorders) | 7 (9) | 10 (13)
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 8 (8) | 14 (14)
Upper respiratory infection (Infections and infestations) | 7 (7) | 7 (8)
Aspartate aminotransferase increased (Investigations) | 6 (9) | 5 (5)
Hypertension (Vascular disorders) | 7 (7) | 5 (6)
Dehydration (Metabolism and nutrition disorders) | 5 (5) | 5 (5)
Cholesterol high (Investigations) | 4 (4) | 3 (5)
Serum amylase increased (Investigations) | 2 (2) | 4 (7)
Thromboembolic event (Vascular disorders) | 4 (6) | 3 (3)
Blood bilirubin increased (Investigations) | 3 (3) | 3 (5)
Vascular access complication (Injury, poisoning and procedural complications) | 3 (4) | 3 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (3) | 2 (4)
Hypokalemia (Metabolism and nutrition disorders) | 2 (4) | 3 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 4 (6)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 2 (3)
Mucosal infection (Infections and infestations) | 2 (3) | 2 (2)
Skin infection (Infections and infestations) | 2 (2) | 2 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 1 (1)
Lipase increased (Investigations) | 1 (1) | 3 (3)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hypotension (Vascular disorders) | 1 (1) | 3 (3)
Fever (General disorders) | 1 (1) | 2 (2)
General disorders and administration site conditions - Other (General disorders) | 0 (0) | 2 (3)
GGT increased (Investigations) | 1 (1) | 2 (2)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Headache (Nervous system disorders) | 1 (1) | 2 (2)
Neuralgia (Nervous system disorders) | 1 (1) | 2 (2)
Peripheral motor neuropathy (Nervous system disorders) | 2 (2) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 2 (2)
Allergic reaction (Immune system disorders) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Syncope (Nervous system disorders) | 0 (0) | 2 (2)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MSA states Site is unable to publish until all completed case report forms have been delivered to Sponsor, (Study Completion). Site shall have the right to publish after publication of a multi-center publication coordinated by the Sponsor or (12) mths. after Study Completion; provided, that prior to any such publication or public release of such data, Site shall furnish Sponsor with a copy of any proposed publication at least (45)days in advance of the proposed publication or presentation date.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-01): https://cdn.clinicaltrials.gov/large-docs/67/NCT04401267/Prot_SAP_001.pdf
  • Informed Consent Form (2021-03-01): https://cdn.clinicaltrials.gov/large-docs/67/NCT04401267/ICF_000.pdf